CLINICAL TRIAL: NCT04098107
Title: A Low-Cost, Collaborative Tool for the Tracking of Youth Activities to Reduce Risk of Physical Injury
Brief Title: Throwing Device Tracker for Youth Injury Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 19-016149; 1R43HD098958-01 (NIH)
Record Dates: First submitted 2019-08-12; First posted 2019-09-23 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Overuse Injury
Keywords: Healthy subjects; Athletes; Baseball; Sports research; overuse injuries
MeSH Terms: conditions — Cumulative Trauma Disorders

STUDY DESIGN:
Intervention Model Description: a wearable prototype device for monitoring upper extremity sports related forces translated to the body during activity. The system will track exposure to injurious forces and monitor adherence to sport specific overuse standards and prescribed rehab regimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Throwing Device Phase 1 (Experimental): During Phase 1, subjects that have been recruited, consented, and enrolled will come to the biomechanics laboratory for throwing performance housed at the University of Pennsylvania (Human Motion Laboratory) on the day of their appointment. Subjects will be asked to wear the prototype device during a simulated baseball game (approximately 30-45 pitches), and then will perform a set of other baseball-specific movements while fitted with infrared markers for throwing analysis. This data will be used to develop and refine the algorithm for the prototype.
  Interventions: Device: Throwing Device

INTERVENTIONS:
Device: Throwing Device — The Innovative Design Labs ( IDL) PhySens will be used to monitor the physical motions of subjects during standard sports-related actions (e.g. throwing a baseball). For this test, the PhySens Carrier will be attached via clothing rivets to a fabric sleeve or strap made of compliant materials commonly used in clothing and wearable products (e.g. nylon, spandex, neoprene).

SUMMARY:
The primary objective of this study is to collect motion-capture data on movements common to baseball play in order to develop an algorithm for a wearable device for the prevention and rehabilitation of sports-related overuse injuries. Secondary objectives include evaluating the feasibility of wearing the throwing device during simulated baseball play.

DETAILED DESCRIPTION:
With the rise in competitive sports participation in pediatric and adolescent populations, there has also been an increase in overuse injuries. Current methods of overuse injury prevention, such as pitch-counting, fail to account for differing techniques or effort and often ignore the elevated risk for children participating in two or more sports emphasizing the same body part. This wearable device seeks to more accurately monitor overuse to prevent and aid rehabilitation of overuse injuries.

Subjects will be asked to fill out a short survey about their athletic activities. They will wear a prototype of a minimal risk throwing device during simulated baseball play in a sports medicine session or at the Human Motion Laboratory. Various motion data from the device and from the Motion Lab analysis will be collected to create and refine an algorithm to quantify workload and throwing movements.

The primary endpoint of this study is to quantify motion capture data on movements common to baseball play. The secondary endpoints include quantifying injury associated with different baseball movement using the proposed system, development of algorithms to quantify workloads associated with injury during common baseball movements and validation of basic device measurements (Pilot Phase).

ELIGIBILITY:
Inclusion Criteria:

Pilot Phase:

1. Males or females age 8 to 14 years
2. Presenting to the Children's Hospital of Philadelphia (CHOP) Physical Therapy Clinic for rehabilitation of injury that does not impede their ability to perform basic throwing movements.

Phase 1:

1. Males or females age 8 to 14 years
2. Involved in official baseball team and primarily plays as the pitcher

Exclusion Criteria:

Pilot Phase

1. Injury of any aspect of the throwing arm
2. Unwillingness to perform all requested motions
3. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study procedures.

Phase 1

1. Injury or disability impeding ability to perform normal baseball-related movements
2. Inability/unwillingness to schedule and/or travel to the Human Motion Laboratory
3. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Greenberg, PT,DPT,PhD, Principal Investigator — Children's Hospital of Philadelphia; J. Todd Lawrence, MD, PhD, Study Director — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Throwing Device Phase 1: 10 patients were recruited
Period: Overall Study
Arm/Group | Throwing Device Phase 1
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Throwing Device Phase 1: Subjects were asked to wear the prototype device during a simulated baseball game (approximately 30-45 pitches), and then perform a set of other baseball-specific movements while fitted with infrared markers for throwing analysis. This information to help us develop a small wearable device that collects and tracks information (such as force) about throwing movements during youth athletic activity to identify and track arm fatigue
Arm/Group | Throwing Device Phase 1
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.3 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race - White | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of the Pitching Detection Algorithm
Description: The number of pitches thrown were tracked and counted visually during data collection. The actual pitch count was then compared to the pitch count logged by the device algorithm to determine the accuracy of the algorithm in detecting pitching events.
Time Frame: 12 months
Population: Our criteria for success was the accuracy of pitching event detection, which was 98.6%
Measure: Number; unit: percentage
Arm/Group | Throwing Device Phase 1
Number analyzed (Participants) | 10
percentage | 98.6

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Clinical adverse events (AEs) will be monitored throughout the study. Since the study procedures are not greater than minimal risk, Serious Adverse Events are not expected.
Arm/Group | Throwing Device Phase 1
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT04098107/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT04098107/ICF_001.pdf